CLINICAL TRIAL: NCT00295555
Title: Effects of Doxazosin on Ambulatory Blood Pressure and Sympathetic Nervous Activity in Hypertensive Patients With Diabetic Nephropathy
Brief Title: Doxazosin Effects on ABPM in Hypertensive Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yokohama City University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7332-2
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus; Essential Hypertension; Renal Failure
Keywords: ambulatory blood pressure monitoring; doxazosin; alpha1-adrenergic antagonists; sympathetic nervous activity; diabetic nephropathy; essential hypertension; power spectral analysis; morning surge
MeSH Terms: conditions — Diabetes Mellitus; Essential Hypertension; Renal Insufficiency; Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Effects of doxazosin on morning surge in diabetic patients

SUMMARY:
Few studies have reported the effect of alpha1-adrenergic antagonists on 24-h blood pressure and regulation of sympathetic nervous activity in hypertensive patients with diabetic nephropathy. Using ambulatory blood pressure monitoring devices equipped with spectral analysis of heart rate variability, we assess the effects of doxazosin on blood pressure in diabetic nephropathy patients and compare the results with those in patients with essential hypertension, patients with diabetes mellitus and patients with chronic nephropathy.

DETAILED DESCRIPTION:
The study is an open-labeled parallel prospective trial comparing the effects of doxazosin (2-8 mg/day) on 24-h blood pressure and autonomic nervous activity. Hypertensive patients with non-insulin-dependent diabetic nephropathy, patients with essential hypertension, patients with diabetes mellitus and patients with chronic nephropathy undergo ambulatory blood pressure monitoring before and after treatment with doxazosin. Simultaneously, spectral analysis is performed to calculate the high frequency components as a marker of parasympathetic nervous activity, and the low frequency components/high frequency components ratios as an index of the sympathovagal balance.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients with diabetes mellitus
* Hypertensive patients
* Hypertensive patients with renal disease

Exclusion Criteria:

* Cardiac, hematologic or hepatic disease
* Renal insufficiency (serum creatinine values> 2 mg/L)
* Hormone-induced hypertension
* Cerebral infarction or hemorrhage
* Other major diseases

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Normalization of high blood pressure | One year

CONTACTS AND LOCATIONS:
Overall Officials: Gen Yasuda, MD, Principal Investigator — Yokohama City University Center Hospital
Locations (1):
- Yokohama City University Center Hospital, Yokohama, Japan

REFERENCES:
- [Background] Yasuda G, Hasegawa K, Kuji T, Ogawa N, Shimura G, Umemura S, Tochikubo O. Effects of doxazosin on ambulatory blood pressure and sympathetic nervous activity in hypertensive Type 2 diabetic patients with overt nephropathy. Diabet Med. 2005 Oct;22(10):1394-400. doi: 10.1111/j.1464-5491.2005.01636.x. PMID 16176202
- [Background] Yasuda G, Ando D, Hirawa N, Umemura S, Tochikubo O. Effects of losartan and amlodipine on urinary albumin excretion and ambulatory blood pressure in hypertensive type 2 diabetic patients with overt nephropathy. Diabetes Care. 2005 Aug;28(8):1862-8. doi: 10.2337/diacare.28.8.1862. PMID 16043724
- [Background] Yasuda G, Hasegawa K, Kuji T, Ogawa N, Shimura G, Umemura S, Tochikubo O. Perindopril effects on ambulatory blood pressure: relation to sympathetic nervous activity in subjects with diabetic nephropathy. Am J Hypertens. 2004 Jan;17(1):14-20. doi: 10.1016/j.amjhyper.2003.08.005. PMID 14700506
- [Derived] Yasuda G, Saka S, Ando D, Hirawa N. Effects of doxazosin as the third agent on morning hypertension and position-related blood pressure changes in diabetic patients with chronic kidney disease. Clin Exp Hypertens. 2015;37(1):75-81. doi: 10.3109/10641963.2014.913599. Epub 2014 May 27. PMID 24866870